CLINICAL TRIAL: NCT06065371
Title: Sacituzumab Govitecan in Combination With Capecitabine for Advanced Gastrointestinal Cancers After Progression on Standard Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Maria Diab, Assistant Professor, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFH-23-03
Record Dates: First submitted 2023-09-13; First posted 2023-10-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer
Keywords: pancreatic cancer; biliary tract cancers; colorectal cancer; esophageal cancer; gastroesophageal cancer; gastric cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Capecitabine; sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: 3+3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sacituzumab govitecan and capecitabine (Experimental): The trial has three dose levels. Dose level -1 has capecitabine at 500mg/m2 twice daily taken orally for two weeks on and one week off, plus sacituzumab govitecan at 7.5mg/kg given intravenously on Days 1 and 8. Each cycle is 21 days. Dose level 0 has capecitabine at 500mg/m2 and sacituzumab govitecan at 10mg/kg. Dose level 1 has capecitabine at 825mg/m2 and sacituzumab govitecan at 10mg/kg.
  Interventions: Drug: Capecitabine; Drug: Sacituzumab govetican

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is a fluoropyrimidine that is metabolized to 5-fluorouracil, which inhibits thymidylate synthase. Capecitabine is available in white or off-white tablets with doses of 500mg and 150mg doses. 500mg dose tablets will be used on this trial. Capecitabine will be ordered as a standard of care and provided commercially.
  Other Names: Xeloda
Drug: Sacituzumab govetican — Sacituzumab govitecan is an antibody-drug conjugate that targets Trop-2-expressing cells and is covalently attached to the topoisomerase I inhibitor SN-38. Sacituzumab govitecan will be provided by Gilead Sciences.
  Sacituzumab govitecan for injection, 180 mg and 200 mg, is available as a powder that is to be reconstituted with 20 mL of 0.9% Sodium Chloride Injection prior to intravenous infusion.
  Following reconstitution, each single-dose vial of Sacituzumab govitecan results in a concentration of 10mg/mL with pH of 6.5.
  Other Names: Trodelvy

SUMMARY:
This is a Phase I study to evaluate the safety and tolerability of sacituzumab govitecan in combination with capecitabine for advanced gastrointestinal cancers after progression on standard therapy, and to assess correlation of outcomes with the biomarker Trop-2.

DETAILED DESCRIPTION:
This is a single institution, open-label phase I trial that aims to assess the safety of combination sacituzumab govitecan plus capecitabine in the treatment of patients with gastrointestinal cancers after progression on standard therapy. Gastrointestinal cancers eligible include pancreaticobiliary cancers, colorectal cancers, and upper gastrointestinal cancers such as esophageal, gastroesophageal junction, and gastric cancers. The trial follows a 3 + 3 design and has three planned dose levels. The starting dose of sacituzumab govitecan is 7.5mg/kg intravenously on Days 1 and 8. The starting dose of capecitabine is 500mg/m2 orally twice daily for two weeks on and one week off. Plan is accrue a total of 20 patients.

The primary endpoint is the recommended phase 2 dose (RP2D) Secondary Endpoints include adverse events, objective response rate (ORR), duration of response (DoR), progression-free survival (PFS), and overall survival (OS), There is an exploratory endpoint of the correlation between Trop-2 expression and clinical outcomes.

Patients will be recruited from the Gastrointestinal (GI) Medical Oncology clinics within the Henry Ford Cancer Institute (HFCI) campuses. The study is divided into a Screening period, Treatment period, End of Treatment (EOT) period, and Follow-up period.

During Screening period patients will provide written informed consent (ICF) to participate in the study before completing any protocol-specified procedures or evaluations not considered to be part of the patient's standard care. Procedures that were performed for standard of care prior to signing informed consent may be used for screening purposes (e.g., full physical exam) as long as the procedures were completed within the 28-day screening period. After signing the ICF, patients will be evaluated for entry criteria during the screening period within 28 days before administration of study drugs. Rescreening after screen failure will be allowed.

Treatment will continue until unacceptable toxicity, death, progression of disease (PD) per RECIST 1.1, Investigator's decision to discontinue treatment, the patient withdraws consent, is lost to follow-up, or Institution decides to terminate the trial. Patients with PD per RECIST 1.1 but with otherwise stable or improved performance and clinical status may continue to be treated in the event of a perceived benefit per Investigator; see Section "Treatment beyond progression". Patients with a partial response (PR) or stable disease (SD) will continue to receive treatment until achievement of a confirmed complete response (CR), disease progression, or intolerance to therapy. It is at the discretion of the Investigator to continue treating patients with a confirmed CR.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, 18 years of age or older, able to understand and give written informed consent
* Patients with the histologically or cytologically documented metastatic adenocarcinoma of gastrointestinal origin, including gastroesophageal, colorectal, and pancreaticobiliary that have failed standard therapy
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3, and platelets ≥ 100,000/μL).
* Adequate hepatic function (bilirubin ≤ 1.5x upper limit normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5xULN or ≤ 5xULN if known liver metastases, and serum albumin > 3 g/dL).
* Adequate renal function (Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation.
* Male and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (total abstinence [if it is her preferred and usual lifestyle], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 6 months after study drug discontinuation. For sites outside of the European Union (EU), it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the subject, then the subject must agree to use a medically acceptable method of contraception, ie, double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide. If currently abstinent, the subject must agree to use a highly effective method as described above if she becomes sexually active during the study period or for 6 months after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 28 days before dosing and must continue to use the same contraceptive during the study and for 6 months after study drug discontinuation.
* Male subjects who are partners of women of childbearing potential must use a condom and spermicide and their female partners, if of childbearing potential, must use a highly effective method of contraception (see methods described above in Inclusion Criterion 15) beginning at least 1 menstrual cycle prior to starting study drug, throughout the entire study period, and for 3 months after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile.
* Willing and able to comply with the requirements and restrictions in this protocol

Exclusion Criteria:

* Positive serum pregnancy test or women who are breastfeeding.
* Known hypersensitivity to the study drug(s), its metabolites, or formulation excipient.
* Requirement for ongoing therapy with or prior use of any prohibited medications listed in protocol.
* Have had a prior anticancer biologic agent within 4 weeks prior to enrolment or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrollment and have not recovered (i.e., ≥ Grade 2 is considered not recovered) from adverse events (AEs) at the time of study entry. Note: patients with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study. Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Have previously received topoisomerase 1 inhibitors.
* Have an active second malignancy. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrolment, or patients with surgically cured tumors with low risk of recurrence (e.g., nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
* Have unstable brain metastases. Note: Patients with stable brain metastasis can be included. "Stable" brain metastases may be defined as: Prior local treatment by radiation, surgery, or stereotactic surgery, imaging - stable or decreasing size after such local treatment, clinically stable signs and symptoms for at least 4 weeks, ≥2 weeks from discontinuation of anti-seizure medication. Patient may receive low and stable doses of corticosteroids ≤ 20 mg prednisone or equivalent daily. It should be confirmed by MRI/CT scan that patient has had stable brain metastasis for 4 weeks prior to treatment.
* Met any of the following criteria for cardiac disease:

  * Myocardial infarction or unstable angina pectoris within 6 months of enrolment.
  * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
  * New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%.
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrolment.
* Have active serious infection requiring antibiotics.
* Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

  * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
  * Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
  * Patients who test positive for HIV antibody.
* Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow- up examinations.
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study [list examples as necessary].
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 18 months
  Recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Adverse Events (AEs) | Through study completion, an average of 18 months
  Measure toxicity using National Cancer Information Center (NCIC) criteria v4.0. Measurement
Objective response rate (ORR) | Through study completion, an average of 18 months
  Cross sectional imaging and RECIST criteria
Duration of Response (DoR) | 18 months
  Time from best response measured by RECIST until progression
Progression-free Survival (PFS) | 18 months
  Survival from starting treatment until progression
Overall Survival (OS) | 18 months
  Survival from starting treatment until death

OTHER OUTCOMES:
Exploratory Endpoint | 18 months
  Correlation between Trop-2 expression and overall response rates and progression-free and overall survivals

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Cancer-Detroit, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Starodub AN, Ocean AJ, Shah MA, Guarino MJ, Picozzi VJ Jr, Vahdat LT, Thomas SS, Govindan SV, Maliakal PP, Wegener WA, Hamburger SA, Sharkey RM, Goldenberg DM. First-in-Human Trial of a Novel Anti-Trop-2 Antibody-SN-38 Conjugate, Sacituzumab Govitecan, for the Treatment of Diverse Metastatic Solid Tumors. Clin Cancer Res. 2015 Sep 1;21(17):3870-8. doi: 10.1158/1078-0432.CCR-14-3321. Epub 2015 May 5. PMID 25944802
- [Background] Fong D, Moser P, Krammel C, Gostner JM, Margreiter R, Mitterer M, Gastl G, Spizzo G. High expression of TROP2 correlates with poor prognosis in pancreatic cancer. Br J Cancer. 2008 Oct 21;99(8):1290-5. doi: 10.1038/sj.bjc.6604677. Epub 2008 Sep 23. PMID 18813308
- [Background] Ohmachi T, Tanaka F, Mimori K, Inoue H, Yanaga K, Mori M. Clinical significance of TROP2 expression in colorectal cancer. Clin Cancer Res. 2006 May 15;12(10):3057-63. doi: 10.1158/1078-0432.CCR-05-1961. PMID 16707602
- [Background] Zhao W, Zhu H, Zhang S, Yong H, Wang W, Zhou Y, Wang B, Wen J, Qiu Z, Ding G, Feng Z, Zhu J. Trop2 is overexpressed in gastric cancer and predicts poor prognosis. Oncotarget. 2016 Feb 2;7(5):6136-45. doi: 10.18632/oncotarget.6733. PMID 26716416
- [Background] Bardia A, Tolaney SM, Punie K, Loirat D, Oliveira M, Kalinsky K, Zelnak A, Aftimos P, Dalenc F, Sardesai S, Hamilton E, Sharma P, Recalde S, Gil EC, Traina T, O'Shaughnessy J, Cortes J, Tsai M, Vahdat L, Dieras V, Carey LA, Rugo HS, Goldenberg DM, Hong Q, Olivo M, Itri LM, Hurvitz SA. Biomarker analyses in the phase III ASCENT study of sacituzumab govitecan versus chemotherapy in patients with metastatic triple-negative breast cancer. Ann Oncol. 2021 Sep;32(9):1148-1156. doi: 10.1016/j.annonc.2021.06.002. Epub 2021 Jun 8. PMID 34116144